CLINICAL TRIAL: NCT05058625
Title: Influence of Latent Miofascial Trigger Points in the Vertical Jump in Female Voleyball Players
Acronym: LMTP_Volley
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sánchez-Sierra1
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — Dry Needling; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needly Group (Experimental): Once the trigger point has been identified, we will use the Hong tecnique looking for a local spasm response
  Interventions: Device: Dry Needling plus normal volleyball training
- Control Group (Active Comparator): Normal volleyball training
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Dry Needling plus normal volleyball training — Once the trigger point has been identified, we will use the Hong tecnique looking for a local spasm response
  Arms: Needly Group
Other: Control Group — Normal volleyball training
  Arms: Control Group

SUMMARY:
To evaluate the effects of dry needling of latent myofascial trigger points on vertical jump height in female volleyball players

DETAILED DESCRIPTION:
Evaluate a sample of female volleyball players after using dry needling on latent myofascial trigger points and verify if it would have an improvement of the vertical jump

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volleyball players
* No Lower limbs injuries in the last 6 months
* Presence of latent trigger points in gastrocnemius
* Familiar with performing CMJ test

Exclusion Criteria:

* Active trigger points in the lower limbs
* Any contraindication of usind dry needling
* Any pathology that prevented the performance of CMJ test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Volleyball Players
Enrollment: 50 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump | pre-intervention
  Vertical jump will be measured CMJ test using the app My Jump 2
Vertical Jump | Immediately post-intervention
  Vertical jump will be measured CMJ test using the app My Jump 2
Vertical Jump | 72 hours post-intervention
  Vertical jump will be measured CMJ test using the app My Jump 2
Vertical Jump | one week post-intervention
  Vertical jump will be measured CMJ test using the app My Jump 2

CONTACTS AND LOCATIONS:
Locations (1):
- Alberto Sánchez Sierra, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No